CLINICAL TRIAL: NCT02463721
Title: Identification of Ascitic Fluid Bacterial Pathogens in Spontaneous Bacterial Peritonitis in Nile Delta and Its Impact on Clinical Outcome of These Patients
Brief Title: Identification of Ascitic Fluid Bacterial Pathogens in Spontaneous Bacterial Peritonitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, PI, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SBP
Record Dates: First submitted 2015-05-27; First posted 2015-06-04 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Primary Bacterial Peritonitis
Keywords: sbp; culture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SBP patients (Other): ascitic fluid culture and microbiological testing for 100 patients with liver cirrhosis and ascites with suspicion of SBP
  Interventions: Other: ascitic fluid culture and microbiological testing

INTERVENTIONS:
Other: ascitic fluid culture and microbiological testing — ascitic fluid culture and microbiological testing for 100 patients with liver cirrhosis and ascites with suspicion of SBP

SUMMARY:
Several studies have pointed out changes in the epidemiology of the causative bacteria in SBP and bacterascites and in their susceptibility to antibiotics. In particular, the development of beta-lactamase enzymes, which confer resistance to clavulanate, or extended spectrum beta-lactamases in Escherichia coli. The potential emergence of enterococci, methicillin-resistant S. aureus, or fluoroquinolone-resistant bacteria, following norfloxacin prophylaxis, is also a cause of concern since they may be associated with a higher risk of therapeutic failure.

The microbial etiology of SBP remains relatively constant; however, the antibiotic resistance rate especially for third-generation cephalosporins (including cefotaxime and ceftazidime), ciprofloxacin, and ofloxacin increased dramatically

DETAILED DESCRIPTION:
Spontaneous bacterial peritonitis (SBP), defined as an infection of ascites in the absence of a contiguous source of infection.

Spontaneous bacterial peritonitis (SBP) is a common and potentially fatal bacterial infection in patients with cirrhosis and ascites, occurring in 10 to 30% of patients, with in-hospital mortality rates ranging from 20 to 30% .

It is secondary to impaired humoral and cellular immune responses that result in indirect intestinal bacterial translocation into the ascitic fluid.

SBP is also associated with a poor long-term prognosis for patients, as mortality rates can reach 50 to 70% at 1 year.

Early diagnosis and early optimal treatment of these infections with appropriate antibiotics and the prevention of hepatorenal syndrome with albumin are required .

Current European and most other international guidelines recommend the use of a third-generation cephalosporin as the first choice, or amoxicillin-clavulanate acid or fluoroquinolones as an alternative choice.

These recommendations are based mainly on clinical trials that were very often conducted a decade or more ago, and on the assumption that E. coli would be involved in nearly half of the cases.

Several studies have pointed out changes in the epidemiology of the causative bacteria in SBP and bacterascites and in their susceptibility to antibiotics. In particular, the development of beta-lactamase enzymes, which confer resistance to clavulanate, or extended spectrum beta-lactamases in Escherichia coli.The potential emergence of enterococci, methicillin-resistant S. aureus, or fluoroquinolone-resistant bacteria, following norfloxacin prophylaxis, is also a cause of concern since they may be associated with a higher risk of therapeutic failure.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis with ascites and suspected to have SBP.
* ascitic fluid PMNL ≥ 250 cells/mm3

Exclusion Criteria:

* ascitic fluid with polymicrobial infections
* patients started empirical antibiotics without prior culture.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
identification of SBP bacterial pathogens through gram stain or other specific stains | 6 months
  identification of SBP bacterial pathogens through gram stain or other specific stains

CONTACTS AND LOCATIONS:
Overall Officials: Sherief Abd-elsalam, lecturer, Principal Investigator — hepatology dept-Tanta; Sally Elnawasany, lecturer, Study Chair — hepatology dept-Tanta; WALAA eLKHALAWANY, lecturer, Study Chair — hepatology dept-Tanta
Locations (1):
- Tanta university hospital, Tanta, Egypt